CLINICAL TRIAL: NCT05859750
Title: A Multicenter, Open-label, Phase II Study of AK104, a PD-1/CTLA-4 Bispecific Antibody, in Combination With Chemotherapy as First-line Treatment in Patients With Locally Advanced Unresectable or Metastatic Pancreatic Cancer
Brief Title: A Study of AK104 With Chemotherapy as First-line Treatment in Patients With Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-217
Record Dates: First submitted 2023-04-14; First posted 2023-05-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- AK104 6mg/kg and AG (Experimental)
  Interventions: Drug: AK104; Drug: Gemcitabine; Drug: Nab-Paclitaxel
- AK104 10mg/kg and AG (Experimental)
  Interventions: Drug: AK104; Drug: Gemcitabine; Drug: Nab-Paclitaxel
- AK104 and mFOLFIRINOX (Experimental)
  Interventions: Drug: AK104; Drug: Oxaliplatin + Irinotecan + 5-Fluorouracil/Leucovorin
- AK104 and NALIRIFOX (Experimental)
  Interventions: Drug: AK104; Drug: Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate

INTERVENTIONS:
Drug: AK104 — AK104 (6mg/kg) on day 1, IV, Q2W
  Arms: AK104 6mg/kg and AG; AK104 and NALIRIFOX; AK104 and mFOLFIRINOX
Drug: AK104 — AK104 (10mg/kg) on day 1, IV, Q2W
  Arms: AK104 10mg/kg and AG; AK104 and NALIRIFOX; AK104 and mFOLFIRINOX
Drug: Gemcitabine — Gemcitabine (1000mg/m2) on days 1, 8 and 15, IV, Q4W
  Arms: AK104 10mg/kg and AG; AK104 6mg/kg and AG
Drug: Nab-Paclitaxel — Nab-Paclitaxel (125mg/m2) on days 1, 8 and 15, IV, Q4W
  Arms: AK104 10mg/kg and AG; AK104 6mg/kg and AG
Drug: Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate — liposomal irinotecan 50 mg/m², oxaliplatin 60 mg/m², leucovorin 400 mg/m², and fluorouracil 2400 mg/m², administered sequentially as a continuous intravenous infusion over 46 h
  Arms: AK104 and NALIRIFOX
Drug: Oxaliplatin + Irinotecan + 5-Fluorouracil/Leucovorin — oxaliplatin, 85 mg/m²; irinotecan, 180 mg/m²; leucovorin, 400 mg/m²; and fluorouracil, 400 mg/m² given as a bolus followed by 2400 mg per square meter given as a 46-hour continuous infusion, every 2 weeks
  Arms: AK104 and mFOLFIRINOX

SUMMARY:
This study is a multicenter, open-label, phase II study to evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activities of AK104，a PD-1/CTLA-4 bispecific antibody, in combination with chemotherapy as first-line therapy in subjects with advanced unresectable or metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily sign a written informed consent form (ICF), which must be signed before the specified study procedures required for the study are performed.
2. Males or females aged ≥ 18 years and ≤ 75 years at the time of signing the ICF.
3. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC).
4. Patients have not received prior systemic therapy for locally advanced or metastatic pancreatic cancer; for patients who have received prior induction chemotherapy, concurrent chemoradiotherapy, or adjuvant/neoadjuvant chemotherapy for curative intent, the time between disease progression and last treatment should be at least 6 months.
5. Patients have at least one measurable tumor lesion per RECIST v1.1; lesions that received radiotherapy are not selected as target lesions, unless the lesion is the only measurable lesion and has unequivocal progression as judged by imaging, it can be considered as a target lesion.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Expected survival ≥ 3 months.
8. Patients who have adequate organ function.
9. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose and agree to take effective contraception measures during the study drug administration and within 120 days after the last dose. Male patients with female partners of childbearing potential must agree to take effective contraception measures during the study drug administration and within 120 days after the last dose.

Exclusion Criteria:

1. Histologically or cytologically confirmed other pathological types, such as acinar cell carcinoma, pancreatic neuroendocrine neoplasms or pancreatoblastoma.
2. Known active or untreated brain metastases, meningeal metastases, spinal cord compression, or leptomeningeal disease.
3. Patients with known germ line BRAC1/2 mutation.
4. Presence of clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring frequent drainage (≥ 1/month).
5. Patients who, in the opinion of the investigator, have symptoms or signs suggestive of clinically unacceptable deterioration of the primary disease at the time of screening.
6. Active malignancies within the past 3 years, with the exception of tumors in this study and cured local tumors.
7. Major surgery other than the diagnosis of pancreatic cancer within 28 days prior to the first dose or major surgery is expected during the study.
8. Pregnant or lactating women.
9. Patients who received any prior treatments targeting the mechanism of tumor immunity.
10. Patients with known contraindications to prescribed chemotherapy regimen (see instructions for specific drug).
11. Patients with known medical history of severe hypersensitivity reactions to other monoclonal antibodies or intravenous gamma globulin.
12. Active autoimmune disease within 2 years prior to the start of study treatmen.
13. Known active pulmonary tuberculosis.
14. Patients with active hepatitis B or active hepatitis C.
15. Known medical history of immunodeficiency or positive HIV test.
16. Patients with active infection.
17. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
18. Concurrent participation in another clinical study, unless it is an observational, non-interventional clinical study or the follow-up period of an interventional study.
19. Any condition that, in the opinion of the Investigator, may result in a risk when receiving the study drug, or would interfere with the evaluation of the study drug or the safety of patients, or the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR is the proportion of subjects with CR or PR based on RECIST v1.1
The number of subjects experiencing adverse events (AEs) | From the subject signs the ICF to 90 days after the last dose of study treatment.
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of AK104 | From first dose of study drug until the 8th cycle (each cycle is 28 days) of study drug administration.
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Minimum observed concentration (Cmin) of AK104 at steady state | From first dose of study drug until the 8th cycle (each cycle is 28 days) of study drug administration.
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Area under the curve (AUC) of AK104 | From first dose of study drug until the 8th cycle (each cycle is 28 days) of study drug administration.
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of study drug until the 8th cycle (each cycle is 28 days) of study drug administration.
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science And Technology, Wuhan, Hubei
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's hospital, Hangzhou, Zhejiang